CLINICAL TRIAL: NCT01002703
Title: Treatment With Lenalidomide, Bendamustine and Prednisone (RBP) in Patients With Relapsed or Refractory Multiple Myeloma After Autologous Stem Cell Transplantation or Conventional Chemotherapy OSHO #077
Brief Title: Treatment With Lenalidomide, Bendamustine and Prednisone (RBP) in Patients With Relapsed or Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Collaborators: Celgene Corporation (Industry); Mundipharma Pte Ltd. (Industry); Amgen (Industry)
Responsible Party: Prof. Dr. med. Dr. h.c. Dietger Niederwieser, University of Leipzig
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBP-01/08; OSHO77
Record Dates: First submitted 2009-10-23; First posted 2009-10-27 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2009-10

CONDITIONS: Multiple Myeloma
Keywords: Lenalidomide; Bendamustine; Multiple Myeloma; Myeloma; Revlimid; Phase I/II; refractory Myeloma; relapsed Myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Lenalidomide; Bendamustine Hydrochloride; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RBP (Experimental): Lenalidomide and Bendamustine and Prednisone
  Interventions: Drug: Lenalidomide, Bendamustine, Prednisone

INTERVENTIONS:
Drug: Lenalidomide, Bendamustine, Prednisone — During the study the first cohort of subjects receive a starting dose of lenalidomide 10mg/d d1-21, bendamustine 60mg/m²/d d1-2 and prednisone 100mg/d d1-4. Escalation steps will include 15, 20 and 25 mg of lenalidomide and 75mg/m² for bendamustine.

SUMMARY:
Define maximum tolerable dose of the combination lenalidomide, bendamustine, prednisone.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age 18 years at the time of signing the informed consent form.
3. Life expectancy of at least 3 months
4. Able to adhere to the study visit schedule and other protocol requirements
5. Relapsed or refractory MM (only first or second relapse) in stage II or III after autologous SCT or conventional chemotherapy (histologically or cytologically proven/ Salmon and Durie criteria) with detectable myeloma protein in blood or urine
6. All previous cancer therapies, including radiation, cytostatic therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study, without corticosteroids therapy.
7. ECOG performance status of £ 2 at study entry (see Appendix 01).
8. Laboratory test results within ranges
9. Females of childbearing potential must agree to contraception or abstinence
10. Disease free of prior malignancies for ³ 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females.
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Patients with contraindications (exclusion criteria) for treatment with lenalidomide, bendamustine and prednisone.
5. Uncontrolled or severe cardiovascular disease, including myocardial infarction within 6 months before study entry, New York Heart Association Class III or IV heart failure, uncontrolled angina or severe uncontrolled ventricular arrhythmias (≥ Lown 3).
6. Use of any other experimental drug or therapy within 28 days of baseline.
7. Known hypersensitivity to thalidomide or purine analogues
8. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
9. Any prior use of lenalidomide or bendamustine in the last six months
10. Concurrent use of other anti-cancer agents or treatments other stated in this treatment plan.
11. Known positive for HIV or infectious hepatitis, type A, B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerable dose (MTD) of lenalidomide in combination with bendamustine and prednisone (RBP) in refractory and relapsed MM stage I/III | 2 month

SECONDARY OUTCOMES:
To determine the safety of lenalidomide, bendamustine and prednisone at MTD | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leipzig, Leipzig, Germany

REFERENCES:
- See also: Related Info — http://osho.uni-leipzig.de/